CLINICAL TRIAL: NCT01478984
Title: Impact of One Stage Compared With Multistaged PCI Complete Revascularization on Clinical Outcome in Multivessel NSTEMI Patients. Smile Trial
Brief Title: Impact of Different Treatment in Multivessel Non ST Elevation Myocardial Infarction (NSTEMI) Patients: One Stage Versus Multistaged Percutaneous Coronary Intervention (PCI)
Acronym: SMILE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMILE
Record Dates: First submitted 2011-11-11; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Non ST Segment Elevation MI and Unstable Angina
Keywords: NSTEMI; PCI; onestage; multistaged
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- one staged PCI (Active Comparator): the patient randomized to this arms complete the myocardial revascularization in one stage PCI, the investigators treat all lesions.
  Interventions: Procedure: One-Stage group
- multistaged PCI (Active Comparator): the patients randomized to this arms in the first stage the investigators treat only the culprit lesion and in second stage the investigators treat the other vessels
  Interventions: Procedure: Multi-Staged group

INTERVENTIONS:
Procedure: One-Stage group — Patients randomized to One-Stage group were completely revascularizated in one time PCI,
  Arms: one staged PCI
Procedure: Multi-Staged group — patients randomized to Multi-Staged group were completely revascularizated in more time PCI, during the same hospitalization
  Arms: multistaged PCI

SUMMARY:
Patients with NSTEMI and multivessel disease will be scheduled to undergo early invasive strategy (PCI within 72 hours) of de novo native coronary artery lesions were considered for recruitment into the study. Inclusion criteria are the following: diagnosis of NSTEMI according to current guidelines presenting with multivessel disease. We will exclude patients with cardiogenic shock at presentation (systolic blood pressure <90 mmHg despite drug therapy), left main coronary disease (>50% diameter stenosis), previous coronary artery bypass grafting (CABG) surgery, patients with Syntax Score >32 and candidated to by-pass surgery (10), severe valvular heart disease and unsuccessful procedures. Procedure success was defined as the achievement of an angiographic residual stenosis of less than 30% and a thrombolysis in myocardial infarction (TIMI) flow grade III after PCI.

Patients randomized to One-Stage group were completely revascularizated in one time PCI, whereas patients randomized to Multi-Staged group were completely revascularizated in more time PCI, during the same hospitalization. Patients received a clopidogrel loading dose of 600 mg before the PCI (for loading dose administered more than 6 h prior to procedure). Post-procedural antiplatelet regimen consisted of aspirin at 100 mg/day indefinitely and clopidogrel 75 mg/day for at least one month.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of NSTEMI
* presenting with multivessel disease

Exclusion Criteria:

* patients with cardiogenic shock at presentation
* left main coronary disease (>50% diameter stenosis)
* previous coronary artery bypass grafting (CABG) surgery
* patients with Syntax Score >32
* candidated to by-pass surgery
* severe valvular heart disease
* unsuccessful procedures

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Major Adverese Cardiac and cerebral Events (MACCE) | 12 months
  Incidence of major adverse cardiac and cerebrovascular events (MACCE) defined as cardiac or non-cardiac death, inhospital death, re-infarction, re-hospitalisation for acute coronary syndrome, repeat coronary revascularization and stroke at 30 days, 6 months and 1 year.
Major Adverese Cardiac and cerebral Events (MACCE) | 30 days
  Incidence of major adverse cardiac and cerebrovascular events (MACCE) defined as cardiac or non-cardiac death, inhospital death, re-infarction, re-hospitalisation for acute coronary syndrome, repeat coronary revascularization and stroke at 30 days, 6 months and 1 year.
MACCE | 6 months
  Incidence of major adverse cardiac and cerebrovascular events (MACCE) defined as cardiac or non-cardiac death, inhospital death, re-infarction, re-hospitalisation for acute coronary syndrome, repeat coronary revascularization and stroke at 30 days, 6 months and 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Rome, Italy

REFERENCES:
- [Derived] Sardella G, Lucisano L, Garbo R, Pennacchi M, Cavallo E, Stio RE, Calcagno S, Ugo F, Boccuzzi G, Fedele F, Mancone M. Single-Staged Compared With Multi-Staged PCI in Multivessel NSTEMI Patients: The SMILE Trial. J Am Coll Cardiol. 2016 Jan 26;67(3):264-72. doi: 10.1016/j.jacc.2015.10.082. PMID 26796390